CLINICAL TRIAL: NCT00688454
Title: C-Control: Efficacy and Safety of Therapy With Rosuvastatin in Statin-Naive and in Statin-Switched Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr med Madeleine Billeter, AstraZeneca AG, Switzerland
Other Study IDs: NIS-CCH-CRE-2007/1
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Hypercholesteremia
Keywords: Hyperlipidemia; Rosuvastatin; Efficacy; tolerability; CRESTOR therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pt with hypercholesteremia: Patients treated with CRESTOR because of hypercholesteremia

SUMMARY:
The study explores efficacy and safety of the lipid-lowering therapy with CRESTOR in statin-naive patients and in patients with previously unsuccessful statin therapy. This study was designed to investigate the dynamic of the lipid parameters and therapy tolerability during 8-10 weeks treatment with CRESTOR

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypercholesteremia who was never treated with statins before
* Patient with hypercholesteremia who was treated with a statin (other then rosuvastatin) but because of its adverse effects/insufficient action was switched to therapy with CRESTOR

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Statin-naive patients and unsuccessfully treated with other (non rosubastatin) statins patients
Sampling Method: Non-Probability Sample
Enrollment: 3392 (Actual)
Dates: Start 2007-02; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
LDL-Cholesterin, HDL-Cholesterin, Triglycerides, Total Cholesterin | 3 visits within 10 weeks

SECONDARY OUTCOMES:
Tolerability of CRESTOR-therapy | 3 visits within 10 weeks